CLINICAL TRIAL: NCT03769168
Title: An Extension Study of Subcutaneous Secukinumab to Evaluate the Long-term Efficacy, Safety and Tolerability up to 4 Years in Patients With Juvenile Idiopathic Arthritis Subtypes of Juvenile Psoriatic Arthritis and Enthesitis Related Arthritis
Brief Title: An Extension Study of Subcutaneous Secukinumab in Patients With Juvenile Psoriatic Arthritis (JPsA) and Enthesitis Related Arthritis (ERA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAIN457F2304E1; 2018-002521-30 (EudraCT Number)
Record Dates: First submitted 2018-11-21; First posted 2018-12-07 (Actual); Results first posted 2025-05-23 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Juvenile Psoriatic Arthritis; Enthesitis Related Arthritis
Keywords: JIA; JPsA; ERA; Secukinumab; ILAR; Juvenile Psoriatic Arthritis; Enthesitis Related Arthritis
MeSH Terms: conditions — Arthritis, Juvenile | interventions — secukinumab

STUDY DESIGN:
Masking Description: Open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1- Secukinumab 75 mg (Experimental): Participants initially received secukinumab 75mg subcutaneously once every four weeks in the extension study. If the signs and symptoms of the participants were not adequately controlled with the 75mg dose, as determined by the investigator, the dose could be escalated to 150mg subcutaneously. For patients weighing 50kg and over, the dose could further be escalated to 300mg subcutaneously every four weeks. The dose escalation from secukinumab 75mg subcutaneously to 300mg subcutaneously was to be implemented in two steps, with the first step being an increase to 150mg subcutaneously, followed by another escalation to 300mg subcutaneously, based on the judgement of the investigator.
  Interventions: Drug: Secukinumab
- Group 2 - Secukinumab 150 mg (Experimental): Participants initially received secukinumab 150mg subcutaneously once every four weeks in the extension study. If the signs and symptoms of the participants were not adequately controlled with the 150mg dose, as determined by the investigator, the dose could be escalated to 300mg subcutaneously.
  Interventions: Drug: Secukinumab

INTERVENTIONS:
Drug: Secukinumab — Secukinumab solution for subcutaneous injections was provided in PFS. Initially, participants continued to receive secukinumab at either 75 mg (in 0.5mL) or 150 mg (in 1mL) every 4 weeks, consistent with their dosage at the Week 100 visit of the core study. The dose could be escalated from 75 mg to 150 mg for patients whose signs and symptoms were not fully controlled, as judged by the investigator, with the current 75 mg dose. Furthermore, the dose could also be escalated to 300 mg every 4 weeks for patients weighing 50kg and over who were currently on the 150 mg dose and whose signs and symptoms were not well-controlled, as judged by the investigator. The dose escalation from secukinumab 75 mg to 300 mg was to be implemented in two steps (first 150 mg and then 300 mg based on the investigator's judgment). At each study treatment time point, one or two subcutaneous injections in the form of PFS were administered.
  Other Names: AIN457

SUMMARY:
Optional open label, roll over extension study to investigate the efficacy and safety of secukinumab treatment in Juvenile Idiopathic Arthritis (JIA) subtypes of Juvenile Psoriatic Arthritis (JPsA) and Enthesitis Related Arthritis (ERA).

DETAILED DESCRIPTION:
This study is an extension of a previous core study (NCT03031782 [CAIN457F2304]) aiming to assess the long-term efficacy, safety, and tolerability of secukinumab treatment in patients who completed the core study and chose to participate in the extension study. The primary objective was to gather comprehensive data on the efficacy and safety of secukinumab over an extended period.

At Week 104 of the core study, all eligible patients could opt to roll over to the extension study and continue receiving secukinumab at either 75 mg or 150 mg, as they were at the Week 100 visit of the core study. The treatment involved subcutaneous injections using pre-filled syringes (PFS). The duration of patient participation could range from a minimum of one year to a maximum of four years, or until one of the following conditions was met: the drug was locally approved, marketed, and reimbursed, secukinumab could be provided free of charge to patients in compliance with local guidelines, or a maximum of 4 years study duration.

During the extension study (starting from Week 108), to maintain a high proportion of clinically meaningful response during the entire duration of the extension study, the dosing options available, at the Investigator's discretion, were as follows:

* The dose could be escalated from 75 mg to 150 mg for patients whose signs and symptoms were not fully controlled with the current dose of 75 mg and might improve with a higher dose as judged by the investigator
* Further, the dose could be escalated to 300 mg for patients weighing 50 kg and over currently on the 150 mg dose whose signs and symptoms were not fully controlled and might improve further with an increase in dose as judged by the investigator
* Dose escalation from secukinumab 75 mg to 300 mg had to be done in two steps (first 150 mg then 300 mg if the patient weighed 50 kg or over and based on the investigator's judgement), also considering the gap between the two escalations to review the response

ELIGIBILITY:
Key Inclusion Criteria:

* Patients had to have participated in the core study CAIN457F2304 and completed the entire treatment period up to and including Week 104.
* Patients had to be deemed by the investigator to benefit from continued secukinumab therapy.

Key Exclusion Criteria:

* Patients with plans for administration of live vaccines during the extension study period were excluded.
* Patients taking any other concomitant biologic immunomodulating agent(s) except secukinumab were excluded.
* Patients who were deemed not to be benefiting from the study treatment based on lack of improvement or worsening of their symptoms were excluded.

Ages: 2 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2019-06-07 (Actual); Primary Completion 2024-11-07 (Actual); Study Completion 2024-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (23):
- United States (3):
  - St Lukes Intermountain Research Center, Boise, Idaho
  - Cincinnati Childrens Hospital, Cincinnati, Ohio
  - Legacy Emanuel Research Hospital Portland, Portland, Oregon
- Belgium (2):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Ghent
- Germany (3):
  - Novartis Investigative Site, Freiburg im Breisgau
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Saint Augustin
- Italy (2):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Krakow, Poland
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Voronezh
  - Novartis Investigative Site, Yekaterinburg
- South Africa (2):
  - Novartis Investigative Site, Panorama, Western Cape
  - Novartis Investigative Site, Cape Town
- Spain (2):
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Valencia
- Turkey (Türkiye) (4):
  - Novartis Investigative Site, Istanbul, Halkali
  - Novartis Investigative Site, Istanbul, TUR
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2607

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited in 24 centers across 9 countries
Pre-assignment Details: One participant enrolled with planned treatment secukinumab 150 mg discontinued the study before receiving study treatment due to physician decision
Groups:
- Group 1- Secukinumab 75 mg: Participants were planned to initially receive secukinumab 75mg subcutaneously once every four weeks. If the signs and symptoms of the participants were not adequately controlled with the 75mg dose, as determined by the investigator, the dose could be escalated to 150mg subcutaneously. For patients weighing 50kg and over, the dose could further be escalated to 300mg subcutaneously every four weeks. The dose escalation from secukinumab 75mg subcutaneously to 300mg subcutaneously was to be implemented in two steps, with the first step being an increase to 150mg subcutaneously, followed by another escalation to 300mg subcutaneously, based on the judgement of the investigator.
- Group 2 - Secukinumab 150 mg: Participants were planned to initially receive secukinumab 150mg subcutaneously once every four weeks. If the signs and symptoms of the participants were not adequately controlled with the 150mg dose, as determined by the investigator, the dose could be escalated to 300mg subcutaneously.
Period: Overall Study
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg
Started | 19 | 36
Secukinumab Escalated to 150 mg (Participants who had their secukinumab dose escalated to 150 mg) | 6 | 0
Secukinumab Escalated to 300 mg (Participants who had their secukinumab dose escalated to 300 mg) | 2 | 14
Treated | 19 | 35
Completed | 10 | 12
Not Completed | 9 | 24
Not completed — Adverse Event | 0 | 1
Not completed — Lack of Efficacy | 2 | 4
Not completed — Post study access to treatment | 3 | 11
Not completed — Physician Decision | 1 | 4
Not completed — Subject Decision | 2 | 4
Not completed — Guardian decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Participants who enrolled in the extension study. One patient enrolled with planned treatment secukinumab150 mg discontinued the study before receiving study treatment. This patient was not included in the analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total
Number analyzed (Participants) | 19 | 35 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 9.5 (3.49) | 14.1 (2.02) | 12.5 (3.40)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 10 | 18
  Male | 11 | 25 | 36
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 33 | 52
  Other | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Juvenile Idiopathic Arthritis American College of Rheumatology (JIA ACR) 30 Response
Description: The JIA ACR response criteria consisted of 6 core criteria:
  * Physician global assessment of disease activity on a 0-100 mm VAS (0=very good and 100=very poor).
  * Parent's or patients' global assessment of overall well-being on a 0-100 mm VAS (0=very well and 100=very poor).
  * Functional ability (CHAQ: Childhood Health Assessment Questionnaire): 30 questions across 8 domains assessing the child's functional abilities. The total score was calculated as the average of the scores for each domain. It ranged from 0 (no disability) to 3 (very severe disability).
  * Number of joints with active arthritis (as per ACR definition), ranging from 0 to 73.
  * Number of joints with limited range of motion, ranging from 0 to 69.
  * Index of inflammation: C-reactive Protein (CRP) levels The JIA ACR 30 response was achieved if 3 of any 6 core set variables improved by at least 30% from baseline of the core study, and no more than 1 variable worsening more than 30%
Time Frame: Baseline of the core study, Week 104 (start of extension study), 116, 128, 140, 156, 180, 208, 232, 260, 284 , 308 and 312. Study week is defined with respect to the core study.
Population: Participants who enrolled in the extension study. One patient enrolled with planned treatment secukinumab150 mg discontinued the study before receiving study treatment. This patient was not included in the analysis. At each time point, only participants with non-missing values were included in the analysis
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- Total Secukinumab Dose: Total participants from Group 1 and Group 2
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Percentage of Participants
  Week 104 | 100 [79.1 to 100] | 100 [87.7 to 100] | 100 [91.7 to 100]
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | 100 [79.1 to 100] | 96.9 [82.0 to 99.8] | 98.9 [88.2 to 99.9]
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | 100 [78.1 to 100] | 100 [86.3 to 100] | 100 [90.9 to 100]
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | 100 [78.1 to 100] | 100 [87.0 to 100] | 100 [91.3 to 100]
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | 94.7 [71.9 to 99.7] | 100 [87.0 to 100] | 98.1 [88.4 to 99.9]
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | 94.7 [71.9 to 99.7] | 97.0 [82.5 to 99.8] | 96.2 [85.7 to 99.3]
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | 100 [78.1 to 100] | 100 [86.3 to 100] | 100 [90.9 to 100]
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | 94.1 [69.2 to 99.7] | 100 [84.5 to 100] | 97.7 [86.5 to 99.9]
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | 92.9 [64.2 to 99.6] | 96.2 [78.4 to 99.8] | 95.0 [81.8 to 99.1]
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | 100 [73.2 to 100] | 95.7 [76.0 to 99.8] | 97.3 [84.2 to 99.9]
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | 100 [69.9 to 100] | 100 [77.1 to 100] | 100 [85.4 to 100]
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | 90.0 [54.1 to 99.5] | 100 [69.9 to 100] | 95.5 [75.1 to 99.8]

2. Secondary Outcome: Percentage of Participants With JIA ACR 50 Response
Description: The JIA ACR response criteria consisted of 6 core criteria:
  * Physician global assessment of disease activity on a 0-100 mm VAS (0=very good and 100=very poor).
  * Parent's or patients' global assessment of overall well-being on a 0-100 mm VAS (0=very well and 100=very poor).
  * Functional ability (CHAQ): 30 questions across 8 domains assessing the child's functional abilities. The total score was calculated as the average of the scores for each domain (0 [no disability] to 3 [very severe disability]).
  * Number of joints with active arthritis (as per ACR definition), ranging from 0 to 73.
  * Number of joints with limited range of motion, ranging from 0 to 69.
  * Index of inflammation: CRP levels The JIA ACR 50 responses were achieved if 3 of any 6 core set variables improved by at least 50% from baseline of the core study, and no more than 1 variable worsening > 30%
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Percentage of participants
  Week 104 | 94.7 [71.9 to 99.7] | 94.3 [79.5 to 99.0] | 94.4 [83.7 to 98.6]
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | 100 [79.1 to 100] | 93.8 [77.8 to 98.9] | 96.1 [85.4 to 99.3]
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | 94.4 [74.2 to 98.7] | 93.5 [77.2 to 98.9] | 93.9 [82.1 to 98.4]
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | 100 [78.1 to 100] | 90.9 [74.5 to 97.6] | 94.1 [82.8 to 98.5]
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | 94.7 [71.9 to 99.7] | 87.9 [70.9 to 96.0] | 90.4 [78.2 to 96.4]
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | 94.7 [71.9 to 99.7] | 93.9 [78.4 to 98.9] | 94.2 [83.1 to 98.5]
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | 100 [78.1 to 100] | 90.3 [73.1 to 97.5] | 93.9 [82.1 to 98.4]
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | 94.1 [69.2 to 99.7] | 96.3 [79.1 to 99.8] | 95.5 [83.3 to 99.2]
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | 92.9 [64.2 to 99.6] | 96.2 [78.4 to 99.8] | 95.0 [81.8 to 99.1]
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | 100 [73.2 to 100] | 95.7 [76.0 to 99.8] | 97.3 [84.2 to 99.9]
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | 100 [69.9 to 100] | 100 [77.1 to 100] | 100 [85.4 to 100]
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | 90.0 [54.1 to 99.5] | 100 [69.9 to 100] | 95.5 [75.1 to 99.8]

3. Secondary Outcome: Percentage of Participants With JIA ACR 70 Response
Description: The JIA ACR response criteria consisted of 6 core criteria:
  * Physician global assessment of disease activity on a 0-100 mm VAS (0=very good and 100=very poor).
  * Parent's or patients' global assessment of overall well-being on a 0-100 mm VAS (0=very well and 100=very poor).
  * Functional ability (CHAQ): 30 questions across 8 domains assessing the child's functional abilities. The total score was calculated as the average of the scores for each domain (0 [no disability] to 3 [very severe disability]).
  * Number of joints with active arthritis (as per ACR definition), ranging from 0 to 73.
  * Number of joints with limited range of motion, ranging from 0 to 69.
  * Index of inflammation: CRP levels The JIA ACR 70 responses were achieved if 3 of any 6 core set variables improved by at least 70%, from baseline of the core study, and no more than 1 variable worsening > 30%
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Percentage of participants
  Week 104 | 94.7 [71.9 to 99.7] | 82.9 [65.7 to 92.8] | 87.0 [74.5 to 94.2]
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | 94.7 [71.9 to 99.7] | 90.6 [73.8 to 97.5] | 92.2 [80.3 to 97.5]
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | 94.4 [70.6 to 99.7] | 90.3 [73.1 to 97.5] | 91.8 [79.5 to 97.4]
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | 88.9 [63.9 to 98.1] | 84.8 [67.3 to 94.3] | 86.3 [73.1 to 93.8]
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | 94.7 [71.9 to 99.7] | 84.8 [67.3 to 94.3] | 88.5 [75.9 to 95.2]
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | 89.5 [65.5 to 98.2] | 81.8 [63.9 to 92.4] | 84.6 [71.4 to 92.7]
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | 94.4 [70.6 to 99.7] | 90.3 [73.1 to 97.5] | 91.8 [79.5 to 97.4]
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | 88.2 [62.3 to 97.9] | 85.2 [65.4 to 95.1] | 86.4 [72.0 to 94.3]
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | 92.9 [64.2 to 99.6] | 96.2 [78.4 to 99.8] | 95.0 [81.8 to 99.1]
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | 100 [73.2 to 100] | 95.7 [76.0 to 99.8] | 97.3 [84.2 to 99.9]
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | 100 [69.9 to 100] | 100 [77.1 to 100] | 100 [85.4 to 100]
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | 90.0 [54.1 to 99.5] | 83.3 [50.9 to 97.1] | 86.4 [64.0 to 96.4]

4. Secondary Outcome: Percentage of Participants With JIA ACR 90 Response
Description: The JIA ACR response criteria consisted of 6 core criteria:
  * Physician global assessment of disease activity on a 0-100 mm VAS (0=very good and 100=very poor).
  * Parent's or patients' global assessment of overall well-being on a 0-100 mm VAS (0=very well and 100=very poor).
  * Functional ability (CHAQ): 30 questions across 8 domains assessing the child's functional abilities. The total score was calculated as the average of the scores for each domain (0 [no disability] to 3 [very severe disability]).
  * Number of joints with active arthritis (as per ACR definition), ranging from 0 to 73.
  * Number of joints with limited range of motion, ranging from 0 to 69.
  * Index of inflammation: CRP levels The JIA ACR 90 responses were achieved if 3 of any 6 core set variables improved by at least 90% from baseline of the core study, and no more than 1 variable worsening > 30%
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Percentage of participants
  Week 104 | 84.2 [59.5 to 95.8] | 74.3 [56.4 to 86.9] | 77.8 [64.1 to 87.5]
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | 73.7 [48.6 to 89.9] | 75.0 [56.2 to 87.9] | 74.5 [60.1 to 85.2]
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | 83.3 [57.7 to 95.6] | 77.4 [58.5 to 89.7] | 79.6 [65.2 to 89.3]
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | 83.3 [57.7 to 95.6] | 72.7 [54.2 to 86.1] | 76.5 [62.2 to 86.8]
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | 73.7 [48.6 to 89.9] | 75.8 [57.4 to 88.3] | 75.0 [60.8 to 85.5]
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | 84.2 [59.5 to 95.8] | 69.7 [51.1 to 83.8] | 75.0 [60.8 to 85.5]
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | 77.8 [51.9 to 92.6] | 71.0 [51.8 to 85.1] | 73.5 [58.7 to 84.6]
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | 76.5 [49.8 to 92.2] | 81.5 [61.3 to 93.0] | 79.5 [64.2 to 89.7]
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | 71.4 [42.0 to 90.4] | 84.6 [64.3 to 95.0] | 80.0 [63.9 to 90.4]
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | 85.7 [56.2 to 97.5] | 95.7 [76.0 to 99.8] | 91.9 [77.0 to 97.9]
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | 91.7 [59.8 to 99.6] | 88.2 [62.3 to 97.9] | 89.7 [71.5 to 97.3]
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | 80.0 [44.2 to 96.5] | 83.3 [50.9 to 97.1] | 81.8 [59.0 to 94.0]

5. Secondary Outcome: Percentage of Participants With JIA ACR 100 Response
Description: The JIA ACR response criteria consisted of 6 core criteria:
  * Physician global assessment of disease activity on a 0-100 mm VAS (0=very good and 100=very poor).
  * Parent's or patients' global assessment of overall well-being on a 0-100 mm VAS (0=very well and 100=very poor).
  * Functional ability (CHAQ): 30 questions across 8 domains assessing the child's functional abilities. The total score was calculated as the average of the scores for each domain (0 [no disability] to 3 [very severe disability]).
  * Number of joints with active arthritis (as per ACR definition), ranging from 0 to 73.
  * Number of joints with limited range of motion, ranging from 0 to 69.
  * Index of inflammation: CRP levels The JIA ACR 100 responses were achieved if 3 of any 6 core set variables improved with 100% from baseline of the core study, and no more than 1 variable worsening > 30%
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Percentage of participants
  Week 104 | 63.2 [38.6 to 82.8] | 57.1 [39.5 to 73.2] | 59.3 [45.1 to 72.1]
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | 63.2 [38.6 to 82.8] | 62.5 [43.7 to 78.3] | 62.7 [48.1 to 75.5]
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | 66.7 [41.2 to 85.6] | 54.8 [36.3 to 72.2] | 59.2 [44.3 to 72.7]
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | 66.7 [41.2 to 85.6] | 57.6 [39.4 to 74.0] | 60.8 [46.1 to 73.8]
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | 63.2 [38.6 to 82.8] | 60.6 [42.2 to 76.6] | 61.5 [47.0 to 74.4]
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | 57.9 [34.0 to 78.9] | 54.5 [36.6 to 71.5] | 55.8 [41.4 to 69.3]
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | 72.2 [46.4 to 89.3] | 58.1 [39.3 to 74.9] | 63.3 [48.3 to 76.2]
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | 58.8 [33.5 to 80.6] | 63.0 [42.5 to 79.9] | 61.4 [45.5 to 75.3]
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | 71.4 [42.0 to 90.4] | 65.4 [44.4 to 82.1] | 67.5 [50.8 to 80.9]
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | 78.6 [48.8 to 94.3] | 78.3 [55.8 to 91.7] | 78.4 [61.3 to 89.6]
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | 91.7 [59.8 to 99.6] | 76.5 [49.8 to 92.2] | 82.8 [63.5 to 93.5]
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | 80.0 [44.2 to 96.5] | 75.0 [42.8 to 93.3] | 77.3 [54.2 to 91.3]

6. Secondary Outcome: Number of Participants With Inactive Disease Status
Description: Inactive disease status was confirmed in a patient when all the following conditions were met:
  * No joints with active arthritis
  * No uveitis
  * CRP value within normal limits for the laboratory where tested or, if elevated, not attributable to JIA
  * Physician's global assessment of disease activity score ≤ 10mm
  * Duration of morning stiffness attributable to JIA lasting ≥15 minutes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Percentage of Participants
  Week 104 | 63.2 [38.6 to 82.8] | 65.7 [47.7 to 80.3] | 64.8 [50.6 to 77.0]
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | 68.4 [43.5 to 86.4] | 71.9 [53.0 to 85.6] | 70.6 [56.0 to 82.1]
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | 66.7 [41.2 to 85.6] | 64.5 [45.4 to 80.2] | 65.3 [50.3 to 77.9]
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | 72.2 [46.4 to 89.3] | 63.6 [45.1 to 79.0] | 66.7 [52.0 to 77.9]
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | 68.4 [43.5 to 86.4] | 72.7 [54.2 to 86.1] | 71.2 [56.7 to 82.5]
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | 68.4 [43.5 to 86.4] | 54.5 [36.6 to 71.5] | 59.6 [45.1 to 72.7]
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | 61.1 [36.1 to 81.7] | 67.7 [48.5 to 82.7] | 65.3 [50.3 to 77.9]
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | 70.6 [44.0 to 88.6] | 66.7 [46.0 to 82.8] | 68.2 [52.3 to 80.9]
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | 71.4 [42.0 to 90.4] | 65.4 [44.4 to 82.1] | 67.5 [50.8 to 80.9]
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | 78.6 [48.8 to 94.3] | 78.3 [55.8 to 91.7] | 78.4 [61.3 to 89.6]
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | 83.3 [50.9 to 97.1] | 82.4 [55.8 to 95.3] | 82.8 [63.5 to 93.5]
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | 70.0 [35.4 to 91.9] | 75.0 [42.8 to 93.3] | 72.7 [49.6 to 88.4]

7. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in JIA ACR Core Component - Physician Global Assessment of Disease Activity
Description: The JIA ACR response criteria consisted of 6 core criteria, one of which was the physician global assessment of disease activity. this assessment was conducted using a 100 mm VAS score, where 0 represented the best disease activity and 100 the worst. The change from baseline of the core study of the physician global assessment of disease activity was measured, with a negative change indicating improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Score on a Scale
  Week 104 | -40.0 (18.39) | -42.2 (20.43) | -41.4 (19.59)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -40.3 (18.42) | -41.1 (20.35) | -40.8 (19.46)
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | -40.4 (18.55) | -41.9 (21.33) | -41.3 (20.17)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -39.0 (16.75) | -42.4 (19.18) | -41.2 (18.26)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -39.7 (17.09) | -40.8 (20.72) | -40.4 (19.50)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -38.5 (18.20) | -38.9 (21.71) | -38.8 (20.31)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -39.0 (17.06) | -41.8 (19.45) | -40.8 (18.48)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -38.4 (18.20) | -42.9 (20.86) | -41.1 (19.78)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -37.6 (28.75) | -45.4 (20.74) | -42.7 (23.78)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -43.6 (18.96) | -42.8 (20.53) | -43.1 (19.68)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -43.8 (18.76) | -40.3 (20.51) | -41.7 (19.53)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -44.2 (26.58) | -47.4 (22.05) | -46.0 (23.67)

8. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in JIA ACR Core Component - Parent's or Patients' Global Assessment of Overall Well-being
Description: The JIA ACR response criteria included six core components, one of which was the parent's or patients' global assessment of overall well-being. This assessment was conducted using a 100 mm VAS score, where 0 represented "very well" and 100 "very poor". The change from baseline of the core study in the parent's or patients' global assessment of overall well-being was measured, with a negative change indicating improvement
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Score on a Scale
  Week 104 | -47.1 (25.90) | -38.6 (27.74) | -41.6 (27.17)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -45.4 (25.70) | -37.7 (26.39) | -40.5 (26.15)
  Week 128: number analyzed (Participants) | 17 | 31 | 48
  Week 128 | -46.8 (25.02) | -39.1 (26.69) | -41.8 (26.11)
  Week 140: number analyzed (Participants) | 18 | 33 | 33
  Week 140 | -41.1 (27.57) | -38.7 (27.06) | -38.7 (27.06)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -46.1 (25.41) | -39.2 (27.15) | -41.8 (26.49)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -45.5 (27.24) | -39.8 (27.48) | -41.9 (27.27)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -47.6 (25.70) | -40.3 (28.13) | -43.0 (27.23)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -39.6 (27.23) | -43.4 (28.20) | -41.9 (27.57)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -44.8 (34.52) | -42.8 (29.31) | -43.5 (30.80)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -51.6 (24.97) | -43.2 (31.23) | -46.4 (28.96)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -49.8 (24.23) | -48.5 (31.93) | -49.1 (28.53)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -48.9 (28.45) | -53.5 (30.31) | -51.4 (28.87)

9. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in JIA ACR Core Component - Functional Ability (CHAQ)
Description: The JIA ACR response criteria included six core components, one of which was the functional ability, measured by the CHAQ. The CHAQ questionnaire consisted of 30 questions across 8 domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and activities. Each domain was scored on a 4-point scale, and the total score was calculated as the average of the scores for each domain. The total score ranged from 0 (no disability) to 3 (very severe disability). The change from baseline of the core study in the CHAQ was measured, with a negative change indicating improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Score on a Scale
  Week 104 | -0.599 (0.5490) | -0.636 (0.5967) | -0.623 (0.5754)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -0.605 (0.5469) | -0.617 (0.5811) | -0.613 (0.5631)
  Week 128: number analyzed (Participants) | 17 | 31 | 48
  Week 128 | -0.647 (0.5196) | -0.685 (0.5570) | -0.672 (0.5388)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -0.590 (0.4809) | -0.648 (0.5638) | -0.627 (0.5318)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -0.645 (0.5275) | -0.644 (0.5763) | -0.644 (0.5537)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -0.658 (0.5541) | -0.625 (0.5779) | -0.637 (0.5641)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -0.667 (0.4832) | -0.625 (0.5293) | -0.640 (0.5082)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -0.610 (0.5411) | -0.681 (0.5825) | -0.653 (0.5615)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -0.741 (0.5035) | -0.649 (0.6205) | -0.681 (0.5773)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -0.777 (0.5052) | -0.652 (0.6329) | -0.699 (0.5837)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -0.865 (0.4811) | -0.794 (0.6311) | -0.823 (0.5655)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -0.888 (0.5050) | -1.000 (0.6077) | -0.949 (0.5532)

10. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in JIA ACR Core Component - Number of Joints With Active Arthritis
Description: The JIA ACR response criteria included six core components, one of which was the number of joints with active arthritis. This was determined using the ACR definition, which identifies active arthritis as any joint with swelling or, in the absence of swelling, limitation of motion accompanied by either pain on motion or tenderness not due to deformity. The active joint count ranged from 0 to 73. The change from baseline of the core study in the number of active joints was measured, with a negative change indicating improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Joints
  Week 104 | -8.4 (11.03) | -6.9 (5.26) | -7.4 (7.72)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -8.4 (11.48) | -6.6 (4.50) | -7.3 (7.79)
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | -8.7 (11.81) | -7.3 (5.35) | -7.8 (8.24)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -8.4 (11.81) | -7.0 (5.44) | -7.5 (8.17)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -8.1 (9.77) | -7.1 (5.61) | -7.5 (7.32)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -8.3 (11.66) | -7.0 (5.69) | -7.5 (8.29)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -7.0 (6.12) | -6.7 (5.38) | -6.8 (5.60)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -7.4 (8.48) | -7.0 (5.68) | -7.1 (6.80)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -7.9 (10.14) | -7.5 (5.57) | -7.7 (7.36)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -8.4 (11.61) | -7.0 (5.57) | -7.5 (8.25)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -8.0 (9.70) | -6.5 (4.52) | -7.1 (7.01)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -8.9 (11.59) | -7.5 (5.14) | -8.1 (8.48)

11. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in JIA ACR Core Component - Number of Joints With Limited Range of Motion
Description: The JIA ACR response criteria included six core components, one of which was the number of joints with limited range of motion. A total of 69 joints were assessed for limitation of motion. The change from baseline of the core study in the number of joints with limited range of motion was measured, with a negative change indicating improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Joints
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Joints
  Week 104 | -5.5 (6.20) | -5.3 (4.23) | -5.4 (4.96)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -5.4 (6.24) | -5.7 (4.19) | -5.6 (4.99)
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | -5.5 (6.41) | -6.0 (4.60) | -5.8 (5.28)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -5.7 (6.31) | -6.0 (4.99) | -5.9 (5.43)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -5.2 (5.68) | -4.3 (8.19) | -4.6 (7.32)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -5.3 (6.37) | -5.5 (4.83) | -5.4 (5.38)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -5.1 (5.61) | -5.3 (3.92) | -5.2 (4.56)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -4.5 (5.42) | -5.6 (3.93) | -5.2 (4.53)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -5.2 (6.47) | -5.9 (3.93) | -5.7 (4.90)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -5.1 (5.72) | -6.0 (3.88) | -5.7 (4.61)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -5.2 (5.46) | -5.8 (3.05) | -5.5 (4.14)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -5.3 (6.77) | -6.3 (3.62) | -5.8 (5.17)

12. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in JIA ACR Core Component - CRP Levels
Description: The JIA ACR response criteria included six core components, one of which was CRP levels, an inflammation biomarker. Serum concentrations of CRP were determined, and the change from baseline of the core study was assessed, with negative changes indicating improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: milligram (mg) / liter (L)
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
milligram (mg) / liter (L)
  Week 104 | -15.238 (38.0680) | -19.788 (36.2920) | -18.187 (36.6322)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -11.201 (40.1619) | -21.795 (37.5991) | -17.848 (38.5218)
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | -15.027 (40.3989) | -21.446 (38.2870) | -19.088 (38.7812)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -15.867 (36.7306) | -21.211 (37.0123) | -19.325 (36.6347)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -13.622 (34.4677) | -21.325 (37.3081) | -18.510 (36.1480)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -16.131 (38.0479) | -20.788 (36.9842) | -19.086 (37.0716)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -16.907 (40.1651) | -20.694 (38.1014) | -19.303 (38.4978)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -15.015 (41.4765) | -20.365 (38.9746) | -18.298 (39.5668)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -18.746 (48.0621) | -20.715 (42.7106) | -20.026 (44.0482)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -19.974 (47.7822) | -15.530 (59.2045) | -17.212 (54.5096)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -21.052 (53.0822) | -21.458 (47.6825) | -21.290 (49.0532)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -25.915 (55.0448) | -27.892 (53.5661) | -26.993 (52.9390)

13. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 of 27-joint Juvenile Arthritis Disease Activity Score (JADAS-27)
Description: The JADAS-27 was used for assessment of disease activity, and it included 4 measures:
  * Physician global assessment of disease activity (VAS range: 0 to 10; where 0=very good and 100=very poor)
  * Parent/participant global assessment of well-being (VAS range: 0 to 10; 0=very well and 100=very poor)
  * Count of joints with active disease (range: 0 to 27; where 0= no disease activity and 27= maximum disease activity)
  * Index of inflammation determined by CRP concentration, calculated as: (CRP (mg/l) -10)/10. Before calculation, CRP values <10 mg/l were converted to 10 and CRP values >110 mg/l were converted to 110. The normalized scale ranged from 0 to 10; where 0= no disease activity and 10= maximum disease activity.
  JADAS-27 score was calculated as the sum of the score of its 4 components, ranging from 0 to 57 where 0= no disease activity and 57= maximum disease activity. The change from baseline of the core study was assessed. A negative change from baseline indicated improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Score on a Scale
  Week 104 | -14.436 (7.2274) | -13.731 (7.4131) | -13.979 (7.2876)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -13.984 (7.9693) | -13.632 (7.0546) | -13.763 (7.3314)
  Week 128: number analyzed (Participants) | 17 | 31 | 48
  Week 128 | -14.478 (7.7217) | -14.277 (7.3964) | -14.348 (7.4314)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -14.050 (7.6609) | -14.104 (7.3246) | -14.085 (7.3683)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -14.027 (6.1256) | -14.158 (7.4052) | -14.111 (6.9032)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -14.235 (7.6622) | -13.737 (7.5190) | -13.919 (7.5002)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -13.501 (5.7531) | -13.869 (7.3790) | -13.734 (6.7665)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -13.064 (6.3732) | -14.669 (7.6410) | -14.049 (7.1443)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -13.454 (8.9326) | -15.096 (7.9790) | -14.521 (8.2484)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -15.358 (7.3767) | -14.445 (8.4302) | -14.791 (7.9550)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -14.437 (6.4218) | -14.647 (8.3114) | -14.560 (7.4623)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -15.310 (8.3332) | -17.122 (8.2219) | -16.298 (8.1255)

14. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 of 71-joint Juvenile Arthritis Disease Activity Score (JADAS-71)
Description: The JADAS-27 was used for assessment of disease activity, and it included 4 measures:
  * Physician global assessment of disease activity (VAS range: 0 to 10; where 0=very good and 100=very poor)
  * Parent/participant global assessment of well-being (VAS range: 0 to 10; 0=very well and 100=very poor)
  * Count of joints with active disease (range: 0 to 71; where 0= no disease activity and 71= maximum disease activity)
  * Index of inflammation determined by CRP concentration, calculated as: (CRP (mg/l) -10)/10. Before calculation, CRP values <10 mg/l were converted to 10 and CRP values >110 mg/l were converted to 110. The normalized scale ranged from 0 to 10; where 0= no disease activity and 10= maximum disease activity.
  JADAS-27 score was calculated as the sum of the score of its 4 components, ranging from 0 to 101 where 0= no disease activity and 101= maximum disease activity. The change from baseline of the core study was assessed. A negative change from baseline indicated improvement.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Score on a Scale
  Week 104 | -17.962 (13.2770) | -16.503 (9.0939) | -17.016 (10.6497)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -17.510 (14.0289) | -16.226 (8.2331) | -16.704 (10.6429)
  Week 128: number analyzed (Participants) | 17 | 31 | 48
  Week 128 | -18.595 (14.2989) | -17.083 (9.1148) | -17.619 (11.0980)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -17.384 (13.8172) | -16.861 (9.0858) | -17.046 (10.8540)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -17.448 (11.6294) | -16.855 (9.1102) | -17.072 (9.9946)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -17.709 (13.9552) | -16.556 (9.4998) | -16.977 (11.2105)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -16.723 (8.8183) | -16.675 (9.0536) | -16.693 (8.8753)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -16.005 (10.7335) | -17.262 (9.3685) | -16.776 (9.8143)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -17.239 (13.8602) | -18.019 (9.7594) | -17.746 (11.1907)
  Week 284: number analyzed (Participants) | 14 | 23 | 37
  Week 284 | -19.144 (13.7107) | -17.141 (10.3338) | -17.899 (11.5806)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -18.520 (12.0126) | -17.000 (9.1449) | -17.629 (10.2499)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -19.810 (14.3124) | -19.622 (9.0748) | -19.707 (11.4427)

15. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in Total Enthesitis Count
Description: The following 16 entheseal sites were assessed for the presence or absence of tenderness (enthesitis) on each side of the body:
  * Anterior Entheses: Greater trochanter of the Femur; Medial condyle of the femur; Lateral condyle of the femur
  * Posterior Entheses: Greater tuberosity of humerus; medial epicondyle of humerus; lateral epicondyle of humerus, Achilles tendon; and calcaneal insertion of the plantar fascia.
  Tenderness on examination was recorded as either present (1) or absent (0) for each of the 16 sites, The total enthesitis count ranged from 0 to 16.
  The change from baseline of the core study was assessed. A negative change from baseline indicated improvement
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Enthesitis count
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Enthesitis count
  Week 104 | -2.5 (2.57) | -2.3 (2.30) | -2.4 (2.37)
  Week 116: number analyzed (Participants) | 19 | 32 | 51
  Week 116 | -2.4 (2.36) | -2.3 (2.50) | -2.4 (2.42)
  Week 128: number analyzed (Participants) | 18 | 31 | 49
  Week 128 | -2.4 (2.43) | -2.3 (1.97) | -2.3 (2.13)
  Week 140: number analyzed (Participants) | 18 | 33 | 51
  Week 140 | -2.5 (2.36) | -2.7 (2.43) | -2.6 (2.38)
  Week 156: number analyzed (Participants) | 19 | 33 | 52
  Week 156 | -2.7 (3.03) | -2.5 (2.36) | -2.2 (2.62)
  Week 180: number analyzed (Participants) | 19 | 33 | 52
  Week 180 | -2.6 (2.59) | -2.5 (2.54) | -2.5 (2.53)
  Week 208: number analyzed (Participants) | 18 | 31 | 49
  Week 208 | -2.4 (2.81) | -2.3 (2.56) | 2.53 (2.63)
  Week 232: number analyzed (Participants) | 17 | 27 | 44
  Week 232 | -2.5 (2.85) | -2.0 (2.28) | -2.2 (2.49)
  Week 260: number analyzed (Participants) | 15 | 26 | 41
  Week 260 | -2.5 (3.54) | -2.0 (1.36) | -2.2 (2.37)
  Week 284: number analyzed (Participants) | 14 | 24 | 38
  Week 284 | -2.9 (3.05) | -2.0 (1.52) | -2.4 (2.21)
  Week 308: number analyzed (Participants) | 12 | 17 | 29
  Week 308 | -3.2 (3.07) | -2.1 (1.25) | -2.5 (2.21)
  Week 312: number analyzed (Participants) | 10 | 12 | 22
  Week 312 | -2.5 (2.32) | -2.1 (1.44) | -2.3 (1.86)

16. Secondary Outcome: Change From Baseline of Core Study CAIN457F2304 in Total Dactylitis Count
Description: The dactylitis count was the number of fingers and toes presenting with swelling and inflammation.
  Swelling and inflammation on examination was recorded as either present (1) or absent (0) for each of the 20 sites, The total dactylitis count ranged from 0 to 20.
  The change from baseline of the core study was assessed. A negative change from baseline indicated improvement
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Dactylitis count
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 18 | 35 | 53
Dactylitis count
  Week 104 | -1.3 (1.94) | -0.4 (1.97) | -0.7 (1.99)
  Week 116: number analyzed (Participants) | 18 | 32 | 50
  Week 116 | -1.5 (2.04) | -0.5 (2.05) | -0.9 (2.08)
  Week 128: number analyzed (Participants) | 17 | 31 | 48
  Week 128 | -1.8 (2.39) | -0.5 (2.23) | -0.9 (2.35)
  Week 140: number analyzed (Participants) | 17 | 33 | 50
  Week 140 | -1.6 (2.42) | -0.6 (2.09) | -1.0 (2.24)
  Week 156: number analyzed (Participants) | 18 | 33 | 51
  Week 156 | -1.6 (2.23) | -0.7 (2.07) | -1.0 (2.15)
  Week 180: number analyzed (Participants) | 18 | 33 | 51
  Week 180 | -1.8 (2.41) | 0.0 (4.15) | -0.6 (3.71)
  Week 208: number analyzed (Participants) | 17 | 31 | 48
  Week 208 | -1.6 (2.42) | -0.3 (0.87) | -0.8 (1.70)
  Week 232: number analyzed (Participants) | 16 | 27 | 43
  Week 232 | -1.5 (2.42) | -0.4 (0.88) | -0.8 (1.70)
  Week 260: number analyzed (Participants) | 14 | 26 | 40
  Week 260 | -1.2 (2.04) | -0.3 (0.84) | -0.6 (1.43)
  Week 284: number analyzed (Participants) | 13 | 24 | 37
  Week 284 | -1.2 (2.13) | -0.3 (0.95) | -0.6 (1.52)
  Week 308: number analyzed (Participants) | 11 | 17 | 28
  Week 308 | -0.9 (1.70) | 0.1 (0.56) | -0.3 (1.22)
  Week 312: number analyzed (Participants) | 9 | 12 | 21
  Week 312 | -1.1 (1.83) | -0.2 (0.39) | -0.6 (1.29)

17. Secondary Outcome: Serum Concentrations of Secukinumab Over Time
Description: Serum concentration of secukinumab over time. Blood samples for pharmacokinetics were taken pre-dose at the scheduled time points.
Time Frame: Pre-dose at Week 128, 140, 156, 180, 208, 232, 260, 284 , 308 and 312. Study week is defined with respect to the core study.
Population: Participants who enrolled in the extension study and received at least one dose of study treatment with quantifiable pharmacokinetic (PK) measurements of secukinumab. Participants with dose escalations were not included in the analysis post up-titration.
Measure: Mean (Standard Deviation); unit: microgram (ug)/milliliter (mL)
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 16 | 26 | 42
microgram (ug)/milliliter (mL)
  Week 128: number analyzed (Participants) | 13 | 26 | 39
  Week 128 | 21.4 (8.57) | 26.4 (9.78) | 24.8 (9.58)
  Week 156: number analyzed (Participants) | 16 | 25 | 42
  Week 156 | 20.8 (8.76) | 26.6 (11.6) | 24.3 (10.8)
  Week 180: number analyzed (Participants) | 12 | 22 | 34
  Week 180 | 21.0 (10.4) | 25.2 (9.28) | 23.7 (9.75)
  Week 208: number analyzed (Participants) | 11 | 18 | 29
  Week 208 | 20.5 (6.82) | 26.7 (11.4) | 24.3 (10.2)
  Week 232: number analyzed (Participants) | 10 | 16 | 26
  Week 232 | 19.7 (7.06) | 24.2 (11.6) | 22.5 (10.2)
  Week 260: number analyzed (Participants) | 9 | 13 | 22
  Week 260 | 16.0 (6.94) | 25.4 (8.99) | 21.5 (9.32)
  Week 284: number analyzed (Participants) | 7 | 10 | 17
  Week 284 | 13.5 (7.99) | 27.5 (7.48) | 21.7 (10.3)
  Week 308: number analyzed (Participants) | 7 | 5 | 12
  Week 308 | 12.5 (5.31) | 27.5 (14.7) | 18.8 (12.4)
  Week 312: number analyzed (Participants) | 6 | 5 | 11
  Week 312 | 14.6 (4.79) | 25.4 (18.5) | 19.5 (13.4)

18. Secondary Outcome: Number of Participants With Treatment-emergent Anti-Drug Antibodies (ADAs) of Secukinumab
Description: Number of participants with treatment-emergent Anti-Drug Antibodies (ADAs) of secukinumab. Blood samples were collected for immunogenicity (anti-AIN457 antibodies) assessments.
Time Frame: From baseline of the core study up to Week 312. Study week is defined with respect to the core study.
Population: Participants who enrolled in the extension study and received at least one dose of study treatment with immunogenicity (anti-AIN457 antibodies) measurements of secukinumab in both the core and extension study
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1- Secukinumab 75 mg | Group 2 - Secukinumab 150 mg | Total Secukinumab Dose
Number analyzed (Participants) | 19 | 35 | 54
Participants | 0 | 6 | 6

ADVERSE EVENTS:
Time Frame: From first dose of secukinumab in the extension study up to 84 days after last dose of secukinumab, assessed up to approximately 4 years
Description: Any sign or symptom during the trial, including those starting after the first dose the extension study, and events present prior to the first dose in the extension study but worsened, and within 84 days after last dose. Analyses were conducted in the safety set (all participants who received at least one dose of study drug). AEs were reported according to the dose the participants were receiving when the AE started. For non-serious AEs, only those with a frequency exceeding 5% are reported.
Groups:
- Any Secukinumab 75 mg: Participants who received secukinumab 75 mg dose at any point during the extension study
- Any Secukinumab 150 mg: Participants who received secukinumab 150 mg dose at any point during the extension study
- Any Secukinumab 300 mg: Participants who received secukinumab 300 mg dose at any point during the extension study
- Any Secukinumab: Participants who received secukinumab, regardless of dose, at any point during the extension study
Arm/Group | Any Secukinumab 75 mg | Any Secukinumab 150 mg | Any Secukinumab 300 mg | Any Secukinumab
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/43 | 0/16 | 0/54
Serious Adverse Events (participants affected / at risk) | 0/19 | 4/43 | 0/16 | 4/54
Other Adverse Events (participants affected / at risk) | 15/19 | 28/43 | 11/16 | 43/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab 75 mg (N=19) | Any Secukinumab 150 mg (N=43) | Any Secukinumab 300 mg (N=16) | Any Secukinumab (N=54)
Crohn's disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Acute sinusitis (Infections and infestations) | 0 | 1 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 1
Urethral haemorrhage (Renal and urinary disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any Secukinumab 75 mg (N=19) | Any Secukinumab 150 mg (N=43) | Any Secukinumab 300 mg (N=16) | Any Secukinumab (N=54)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Familial mediterranean fever (Congenital, familial and genetic disorders) | 1 | 0 | 0 | 1
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 1
Astigmatism (Eye disorders) | 0 | 0 | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 0 | 6
Colitis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 5 | 1 | 7
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 3
Vomiting (Gastrointestinal disorders) | 1 | 2 | 0 | 3
Gait disturbance (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 3 | 0 | 3
Swelling face (General disorders) | 1 | 0 | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 1 | 0 | 2
Bacterial infection (Infections and infestations) | 0 | 0 | 1 | 1
Bronchitis (Infections and infestations) | 1 | 2 | 0 | 3
COVID-19 (Infections and infestations) | 1 | 9 | 3 | 13
Cystitis (Infections and infestations) | 0 | 1 | 1 | 1
Ear infection (Infections and infestations) | 0 | 0 | 1 | 1
Eye infection (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 4 | 0 | 4
Gastrointestinal infection (Infections and infestations) | 0 | 1 | 1 | 2
Herpes simplex (Infections and infestations) | 1 | 0 | 0 | 1
Influenza (Infections and infestations) | 1 | 1 | 0 | 2
Nasopharyngitis (Infections and infestations) | 2 | 8 | 4 | 13
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 4 | 0 | 4
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Rhinitis (Infections and infestations) | 1 | 1 | 0 | 2
Sinusitis (Infections and infestations) | 2 | 2 | 1 | 5
Tinea pedis (Infections and infestations) | 1 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 3 | 1 | 4
Tooth abscess (Infections and infestations) | 1 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 2 | 5 | 0 | 7
Vaccination site cellulitis (Infections and infestations) | 1 | 0 | 0 | 1
Varicella (Infections and infestations) | 1 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 4
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 2 | 3
Bacterial test positive (Investigations) | 0 | 0 | 1 | 1
Basophil count increased (Investigations) | 0 | 0 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 1
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 1 | 1
Blood phosphorus increased (Investigations) | 0 | 0 | 1 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 1 | 1
Crystal urine present (Investigations) | 0 | 0 | 1 | 1
Eosinophil count increased (Investigations) | 0 | 0 | 2 | 2
Eosinophil percentage increased (Investigations) | 0 | 0 | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1
High density lipoprotein decreased (Investigations) | 0 | 0 | 1 | 1
Protein urine present (Investigations) | 1 | 0 | 0 | 1
Body fat disorder (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Folate deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Amplified musculoskeletal pain syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7 | 3 | 11
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0 | 5
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 2
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 2
Juvenile idiopathic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3 | 0 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 8 | 0 | 8
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Temporomandibular pain and dysfunction syndrome (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Osteochondroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Headache (Nervous system disorders) | 0 | 3 | 1 | 4
Syncope (Nervous system disorders) | 1 | 1 | 0 | 2
Generalised anxiety disorder (Psychiatric disorders) | 0 | 0 | 1 | 1
Haematuria (Renal and urinary disorders) | 1 | 1 | 0 | 2
Urinary incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 4
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of pooled data (i.e.,data from all sites) in clinical trial or disclosure of trial results in their entirety.

DOCUMENTS (2):
  • Study Protocol (2018-11-12): https://cdn.clinicaltrials.gov/large-docs/68/NCT03769168/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT03769168/SAP_001.pdf